CLINICAL TRIAL: NCT07287228
Title: An Ib/II Phase Clinical Study Evaluating the Safety and Preliminary Efficacy of Daratumumab in Patients With Refractory Aplastic Anemia
Brief Title: The Safety and Efficacy of Daratumumab in Patients With Refractory Aplastic Anemia
Acronym: DARA-AA-001
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Principal Investigator, Jun Shi, Director of the Red Blood Cell Diseases Center & Director of the Regenerative Medicine Clinic, Institute of Hematology & Blood Diseases Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2025084
Record Dates: First submitted 2025-09-25; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Aplastic Anemia; Refractory; Relapse
Keywords: Aplastic anemia, Daratumumab
MeSH Terms: conditions — Anemia, Aplastic; Recurrence | interventions — daratumumab

STUDY DESIGN:
Intervention Model Description: The target population is adult patients with refractory aplastic anemia (AA).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- After enrollment, patients will receive daratumumab treatment. (Experimental): This study is designed as a seamless Phase Ib/II trial. The target population is adult patients with refractory aplastic anemia (AA), who must meet the criteria for refractory AA at enrollment. After enrollment, patients will receive daratumumab treatment.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — In Phase I, eligible subjects who meet the inclusion criteria will receive daratumumab at doses of 8 mg/kg, 12 mg/kg, or 16 mg/kg. The treatment period will last 6 weeks, with intravenous infusion administered once weekly (QW) for a total of 6 consecutive doses.
  During the conduct of the clinical trial, based on the clinical trial data obtained (safety, MTD, etc.) and after discussion by the SRC, the RP2D for Phase II will be determined. In Phase II, eligible subjects who meet the inclusion criteria will receive intravenous daratumumab once weekly (specific dose based on the RP2D determined from Phase Ib clinical trial data after SRC discussion) for a total of 6 consecutive doses.

SUMMARY:
This study consists of two phases, phase Ib and phase II. The primary objective of phase Ib is to evaluate the safety and tolerability of multiple doses of daratumumab in patients with refractory aplastic anemia. The primary objective of phase II is to preliminarily assess the efficacy of multiple doses of daratumumab in patients with refractory aplastic anemia. Secondary objectives include evaluation of other efficacy endpoints, safety (phase II), and pharmacodynamic characteristics of multiple doses of daratumumab in these patients. The exploratory objective is to assess biological functional changes in peripheral blood and bone marrow before and after daratumumab treatment.

DETAILED DESCRIPTION:
This study is a seamless phase Ib/II design. The target population comprises adult patients with refractory aplastic anemia (AA) who meet the criteria for refractory AA at enrollment, with platelet counts (PLT) < 30×10⁹/L or hemoglobin (HGB) < 90 g/L. A Safety Review Committee (SRC), led by the principal investigator, will be established. If the phase Ib results demonstrate sufficient safety and allow determination of the maximum tolerated dose (MTD), the phase II study will proceed directly.

The phase Ib study serves as the dose-escalation stage, with three dose cohorts: low-dose (8 mg/kg), medium-dose (12 mg/kg), and high-dose (16 mg/kg), administered once weekly for six consecutive doses. Dose escalation follows the "3+3" design.

ELIGIBILITY:
Inclusion Criteria:

1. Clearly diagnosed with primary acquired aplastic anemia according to the Chinese Guidelines for the Diagnosis and Treatment of Aplastic Anemia (2022 Edition).
2. Refractory aplastic anemia meeting one of the following criteria:

   2.1 Patients previously diagnosed with severe aplastic anemia (SAA) # or transfusion-dependent non-severe aplastic anemia (TD-NSAA) &: have received antithymocyte/antilymphocyte globulin (ATG/ALG) combined with standard-dose cyclosporine for at least 6 months, and standard-dose thrombopoietin (TPO) receptor agonist* therapy for at least 4 months, but showed no response or relapsed; 2.2 Patients previously diagnosed with non-transfusion-dependent non-severe aplastic anemia (NTD-NSAA): have received standard-dose cyclosporine for at least 6 months, and standard-dose thrombopoietin (TPO) receptor agonist* therapy for at least 4 months, but showed no response or relapsed.
3. Hemoglobin <90 g/L or platelet count <30×10⁹/L.
4. Not suitable for or unwilling to undergo hematopoietic stem cell transplantation; no other better treatment options available.
5. Age ≥18 years, no sex limitation.
6. Eastern Cooperative Oncology Group (ECOG) performance status score ≤2 (see Appendix 2).
7. Voluntarily signed the informed consent form, understands the nature, purpose, and procedures of the trial, and is willing to comply with the trial requirements.

Exclusion Criteria:

1. Patients with congenital bone marrow failure syndromes.
2. Patients with bone marrow reticulin staining ≥ Grade 2.
3. Patients with paroxysmal nocturnal hemoglobinuria (PNH) clone ≥50% or with active hemolysis.
4. Patients with clonal chromosomal abnormalities characteristic of myelodysplastic syndrome (MDS) (except +8, 20q-, and -Y).
5. Presence of active bacterial, viral, or fungal infection within 2 weeks prior to the first administration of the investigational drug (excluding common cold and onychomycosis), or any other severe infection. Any anti-infective therapy for infections must be completed at least 2 weeks before the first dose. History of HIV infection or HIV antibody positive during screening; positive treponema pallidum antibody during screening; active pulmonary tuberculosis (evidenced by chest imaging or other relevant examinations within 3 months prior to first administration or during screening indicating active TB infection); active hepatitis during screening (positive hepatitis B surface antigen [HBsAg], or positive hepatitis B core antibody [HBcAb] with HBV DNA ≥30 IU/mL, or positive hepatitis C antibody [HCV Ab] with positive HCV RNA).
6. Presence of active bleeding in the gastrointestinal tract, respiratory tract, central nervous system, or other sites.
7. History of significant clinical diseases that, in the investigator's judgment, would pose a safety risk for the subject's participation or affect the evaluation of efficacy or safety if the disease/condition worsens during the study. Examples include:

   7.1 Cardiovascular disease: acute myocardial infarction or unstable angina within the past year, severe arrhythmias (such as frequent multifocal PVCs, ventricular tachycardia, ventricular fibrillation, etc.), congestive heart failure, arterial or venous thrombosis, NYHA Class III-IV cardiac function.

   7.2 History of psychiatric disorders or severe cerebrovascular disease or cognitive sequelae.
8. Use of B-cell or plasma-cell targeting agents within 3 months prior to the first administration of the investigational drug or expected use during the study period.
9. Receipt of antithymocyte globulin or antilymphocyte globulin within 6 months prior to the first administration of the investigational drug.
10. Treatment with tacrolimus, sirolimus, cyclophosphamide, anti-CD52 monoclonal antibodies, or similar agents within 4 weeks or 5 half-lives (whichever is shorter) prior to the first administration of the investigational drug.
11. Planned participation in another clinical trial or prior exposure to another investigational product within less than 4 weeks or 5 half-lives (whichever is shorter) before the first dose.
12. Vaccination with live attenuated vaccines within 4 weeks prior to the first administration of the investigational drug or planned during the study period, or COVID-19 vaccination within 7 days prior to first administration.
13. Prior exposure to CD38-targeted therapy.
14. Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study; female subjects of childbearing potential and male subjects with partners of childbearing potential who are unwilling to use highly effective contraception (see Appendix 3 for specific methods) throughout the study (from signing the ICF to 6 months after the last dose of study drug), or who plan to donate eggs or sperm during the study.
15. Any other conditions deemed unsuitable for participation in this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | Within 12 weeks after treatment
  Percentage of patients with hematological response, including complete response (CR) or partial response (PR). Hematological response is evaluated by hemoglobin (Hb), platelet count (PLT) and absolute neutrophil count (ANC).

SECONDARY OUTCOMES:
Incidence of adverse events | Within 12 weeks after treatment
  Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event Use Common Terminology Criteria for Adverse Events (CTCAE) Version 5 to assess the adverse event

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hosptial, Chinese Academy of Medical Science and Peking Union Medical School, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided